CLINICAL TRIAL: NCT04073836
Title: Early Detection of the Cerebral Palsy in Moderate and Late Preterms Through the General Movements
Brief Title: GMA and Peri in Moderate-late Preterms
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Castilla-La Mancha (Other)
Responsible Party: Sponsor
Other Study IDs: jma001
Record Dates: First submitted 2019-08-21; First posted 2019-08-29 (Actual); Last update posted 2019-08-29 (Actual); Status verified 2019-08

CONDITIONS: Preterm; Assessment; Risk Factor; Cerebral Palsy
MeSH Terms: conditions — Premature Birth; Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To analyze the relationship between the early diagnosis of cerebral palsy with the risk factors of this pathology in moderate and late premature infants

DETAILED DESCRIPTION:
Analyze a sample of moderate and late premature infants using general movements and verify which of them would have an early diagnosis of cerebral palsy and relate it to their risk factors for this pathology.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who were born between the week 32 + 0 days and the week 36 + 6 days and who are admitted to the Hospital Nuestra Señora del Prado de Talavera de la Reina or the Hospital Virgen de la Salud de Toledo.

Exclusion Criteria:

* Any type of pre and perinatal diagnostic neurological involvement.
* Any type of pathology associated with prematurity.
* Children who have prescribed any of the following medications (10):

  * Barbiturates
  * Antiepileptic
  * Indomethacin
  * Dexamethasone

Ages: 32 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Subjects who were born between the week 32 + 0 days and the week 36 + 6 days
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
gestation weeks | From date of Recruiting until the discharging of neonatal intensive care unit, assessed up to 40 weeks
  Premature birth week
weight | From date of Recruiting until the discharging of neonatal intensive care unit, assessed up to 40 weeks
  measurement, World Health Organization percentile
size | From date of Recruiting until the discharging of neonatal intensive care unit, assessed up to 40 weeks
  measurement, World Health Organization percentile
cranial perimeter | From date of Recruiting until the discharging of neonatal intensive care unit, assessed up to 40 weeks
  measurement about head, World Health Organization percentile
Apgar | at birth of each preterm
  Outcome about Apgar Test
Magnetic resonance imaging rating scale | From date of Recruiting until the discharging of neonatal intensive care unit, assessed up to 40 weeks
  Outcome about Neuroimaging in preterms
general movements outcome | From date of Recruiting until the discharging of neonatal intensive care unit, assessed up to 40 weeks
  Outcome about General Movements Assessment. Three outcomes about movement of preterm. Normal, Poor Repertoire and Cramped Synchronized
PERI outcome | through study completion, an average of 18 months
  Outcome about Perinatal Risk Scale Scale. Minimum score: 0. Maximum score: 51

CONTACTS AND LOCATIONS:
Locations (1):
- Javier Merino Andrés, Toledo, Spain

IPD SHARING:
Plan to Share IPD: No